CLINICAL TRIAL: NCT03259906
Title: Comparison of Functional Recovery After Distal Intra-articular Radius Fracture With a Dorsal Tilt Treated With an Anterior Plate Versus a Posterior Plate
Acronym: PAPPO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of performance
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALVERNHE LABATTUT 2016
Record Dates: First submitted 2017-08-21; First posted 2017-08-24 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Distal Intra-articular Radius Fracture With a Dorsal Tilt
MeSH Terms: interventions — X-Rays

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Osteosynthesis using a posterior plate (Active Comparator)
  Interventions: Other: DASH score; Procedure: X-ray; Procedure: posterior osteosynthesis
- Osteosynthesis using an anterior plate (Active Comparator)
  Interventions: Other: DASH score; Procedure: X-ray; Procedure: Anterior osteosynthesis

INTERVENTIONS:
Other: DASH score — Questionnaire asking about Disability of Arm, Shoulder and Hand
Procedure: X-ray — postoperative x-rays at 6 weeks, 3, 6 and 12 months
Procedure: posterior osteosynthesis — Osteosynthesis using a posterior plate
  Arms: Osteosynthesis using a posterior plate
Procedure: Anterior osteosynthesis — Osteosynthesis using an anterior plate
  Arms: Osteosynthesis using an anterior plate

SUMMARY:
For les intra-articular fractures, plate osteosynthesis is the indicated technique. Despite the absence of consensus, in recent years, the use of open reduction associated with internal plate fixation has considerably developed. Indeed, this therapeutic option allows a more anatomical reduction and stable fixation.

First-generation posterior plates presented complications related to the size of the plate, notably tendon lesions. Over the last ten years, a new generation of thinner anterior plates has reduced these complications.

In the literature, few studies have compared these two techniques in terms of functional and radiological outcomes. The hypothesis of this research is that osteosynthesis using a posterior plate is more effective than that with an anterior plate in terms of functional recovery in patients older than 45 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have provided written informed consent
* Patients older than 45 years
* Patients presenting a closed intra-articular fracture of the distal radius with a dorsal tilt (stages B2, C1, C2 and C3)

Exclusion Criteria:

* Adults under guardianship
* Patients without national health insurance cover
* Pregnant or breast-feeding women
* Patients presenting other injuries in the same upper limb
* Patients presenting injuries of the wrist or hand (scapholunate injury, fracture of the carpal bone or fingers)
* Pre-trauma paralysis of the limb
* Open fracture
* Fracture with palmer tilt or extra-articular

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-07-04 (Actual); Study Completion 2018-07-04 (Actual)

PRIMARY OUTCOMES:
Evaluation of functional recovery using the DASH questionnaire | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

IPD SHARING:
Plan to Share IPD: Undecided